CLINICAL TRIAL: NCT04037904
Title: Long-term Follow-up of Interleukin-1B and H+,K+-ATPase mRNA Expression After Helicobacter Pylori Eradication
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1509/316-302
Record Dates: First submitted 2019-07-28; First posted 2019-07-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Interleukin-1 beta; Gastric H+, K+- APTase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- H. pylori negative group: Subjects who have not have H. pylori infection, and had not receive H. pylori eradication
- H. pylorieradicated group: Subjects who have had H. pylori infection currently and received successful H. pylori eradication according to appropriated indication

SUMMARY:
We will evaluate the long-term changes of gastric H+, K+-adenosine triphosphatase (H+, K+-ATPase) and Interleukin-1B mRNA expression according to Helicobacter pylori (H.pylori) infection and intestinal metaplasia and investigate the long-term effect of H. pylori eradication

DETAILED DESCRIPTION:
H. pylori suppresses gastric acid secretion by repressing gastric acid pump, H+, K+-ATPase, and stimulating Interleukin-1B. In this study, we will evaluate the expression of H+, K+-ATPase and Interleukin-1B mRNA according to H. pylori infection and intestinal metaplasia in controls and patients with gastric cancer. In addition, we observe the changes of H+, K+-ATPase and Interleukin-1B mRNA expression over 5 years after H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Controls who did not have any evidence of gastric cancer, gastric dysplasia, esophageal tumor, peptic ulcer and lymphoma on esophagogastroduodenoscopy
* Patients with gastric dysplasia or gastric cancer who diagnosed with gastric dysplasia or early gastric cancer in the final pathological report

Exclusion Criteria:

* Subjects with previous eradication treatment for H. pylori
* Subjects with previous gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Controls and patients with gastric dysplasia or gastric cancer who received esophagogastroduodenoscopy and underwent H. pylori tests
Sampling Method: Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Interleukin-1B and H+,K+-ATPase mRNA expression | 1 year
  Gastric Interleukin-1B and H+,K+-ATPase mRNA expression in subjects with and without H. pylori infection at baseline, and changes of Interleukin-1B and H+,K+-ATPase mRNA expression with time in subjects without H. pylori infection and subjects who underwent H. pylori eradication successfully.
  Gastric Interleukin-1B and H+,K+-ATPase mRNA expression measured by reverse transcription polymerase chain reaction, using the gastric mucosa specimen obtained during esophagogastroduodenoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided